CLINICAL TRIAL: NCT05762393
Title: A Phase 1b, Multicenter, Randomized, Placebo-controlled, Observer-blinded, Dose-escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity of the Sm-p80 + GLA-SE (SchistoShield®) Candidate Vaccine in Healthy Adults in Burkina Faso and Madagascar
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of the Sm-p80 + GLA-SE (SchistoShield®) Candidate Vaccine in Healthy Adults in Burkina Faso and Madagascar
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: IVI VASA 001
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Schistosomiasis
Keywords: Vaccine; Schistosomiasis
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The PI, study staff, and participants will be blinded as to receipt of study vaccine or placebo. The unblinded pharmacy staff preparing the study product syringes and the unblinded study nurse who is administering the product will not be involved in the safety assessment of participants and will be instructed not to comment on the experimental agent to study staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Cohort A will receive the low-dose antigen formulation(10 μg Sm-p80 + 5 μg GLA-SE) or placebo. Cohort will include 20 participants randomized to receive either Sm-p80 product or placebo in a 3:1 ratio. All participants will receive three intramuscular injections of 0.5 mL of the designated study product / placebo, on Days 0, 28, and 56 (28 days apart).
  Interventions: Biological: Sm-p80 + GLA-SE
- Cohort B (Experimental): Cohort B will receive the low-dose antigen formulation(30 μg Sm-p80 + 5 μg GLA-SE) or placebo. Cohort will include 20 participants randomized to receive either Sm-p80 product or placebo in a 3:1 ratio. All participants will receive three intramuscular injections of 0.5 mL of the designated study product / placebo, on Days 0, 28, and 56 (28 days apart).
  Interventions: Biological: Sm-p80 + GLA-SE
- Cohort C (Experimental): Cohort C will receive the low-dose antigen formulation(100 μg Sm-p80 + 5 μg GLA-SE) or placebo. Cohort will include 20 participants randomized to receive either Sm-p80 product or placebo in a 3:1 ratio. All participants will receive three intramuscular injections of 0.5 mL of the designated study product / placebo, on Days 0, 28, and 56 (28 days apart).
  Interventions: Biological: Sm-p80 + GLA-SE

INTERVENTIONS:
Biological: Sm-p80 + GLA-SE — Combination vaccine containing Sm-p80 antigen and GLA-SE adjuvant.

SUMMARY:
The goal of this phase 1b, multicenter, randomized, placebo-controlled, observer-blinded, dose-escalation study is to assess the safety, tolerability, and immunogenicity of a three-dose regimen, spaced four weeks apart, given intramuscularly in healthy adults (20-59 years old). Three different dose formulations of the study product with varying antigen contents will be investigated.

A total of 120 eligible participants will be recruited in 3 sequential cohorts (A, B, and C) in Burkina Faso (N=60) and in Madagascar (N=60). Cohort A will receive the low-dose antigen formulation (10 µg) or placebo, Cohort B will receive the medium-dose antigen formulation (30 µg) or placebo, and Cohort C will receive the high-dose antigen formulation (100 µg) or placebo; all antigens with 5 μg adjuvant (GLA-SE). In each cohort, volunteers will be randomized in a blinded manner into one of two arms, candidate vaccine or placebo, by a 3:1 ratio. A subset of five out of 20 subjects in each cohort will be sampled by convenience to enable us to further characterize the immune response using the peripheral blood mononuclear cells (PBMC). The Primary Objective of the study is to evaluate the safety and tolerability of 3 different dose formulations (low dose, medium dose, and high dose) of SchistoShield® vaccine given intramuscularly on D0, D28 and D56 to healthy participants 2018 to 59 years of age in Burkina Faso and Madagascar.

DETAILED DESCRIPTION:
This is a phase 1b, multicenter, randomized, placebo-controlled, observer-blinded, dose-escalation study, assessing the safety, tolerability, and immunogenicity of a three-dose regimen, spaced four weeks apart, given intramuscularly in healthy adults (20-59 years old). Three different dose formulations of the study product with varying antigen contents will be investigated. A total of 120 eligible participants will be recruited in 3 sequential cohorts (A, B, and C) in Burkina Faso (N=60) and in Madagascar (N=60), as shown in the Table 1, below. Cohort A will receive the low-dose antigen formulation (10 µg) or placebo, Cohort B will receive the medium-dose antigen formulation (30 µg) or placebo, and Cohort C will receive the high-dose antigen formulation (100 µg) or placebo; all antigens with 5 μg adjuvant (GLA-SE). In each cohort, volunteers will be randomized in a blinded manner into one of two arms, candidate vaccine or placebo, by a 3:1 ratio. A subset of five out of 20 subjects in each cohort will be sampled by convenience to enable us to further characterize the immune response using the peripheral blood mononuclear cells (PBMC).

To ensure that the study participants at enrollment do not have any active schistosomiasis or helminth infection and are schistosomiasis egg-negative, pre-screening activities including schistosomiasis treatment will be carried out in potential study participants prior to enrollment. Potential study participants will be identified in the catchment population and will be offered anti-helminth treatment using praziquantel (PZQ) and Albendazole (ABZ) as per local guidelines at study site. The pre-screening visit will be conducted 6-8 weeks before the screening visit. The last dose of PZQ/ABZ will be administered at least 5 weeks prior to the first dose of study product.

The Primary objective is to evaluate the safety and tolerability of 3 different dose formulations (low dose, medium dose, and high dose) of SchistoShield® vaccine given intramuscularly on D0, D28 and D56 to healthy participants 20 to 59 years of age in Burkina Faso and Madagascar.

The Secondary objective is to evaluate the immunogenicity of 3 different dose formulations (low dose, medium dose, and high dose) of SchistoShield® vaccine 28 days post-vaccination on D28, D56, and D84 as compared with the baseline and with those who received placebo.

The Exploratory objective is to describe the antigen-specific B- and T-cell responses, memory responses, and innate and adaptive immune signatures from samples collected at specified timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants aged 20 to 59 years at the time of consent.
2. Participant who has completed the deworming using praziquantel (PZQ) and albendazole (ABZ) according to local guidelines, with the last dose of PZQ/ABZ administered at least 5 weeks prior to first dose of study product.
3. Participant who, after the nature of the study has been explained, has voluntarily given informed consent, according to the local regulatory requirements, prior to study entry.
4. Participant who can comply with the study procedures and available for the entire duration of the study (32 weeks).
5. Individuals in good health as determined by the outcome of medical history, physical examination, hematology and biochemistry tests at the time of screening and the clinical judgment of the investigator.
6. Women of childbearing potential* with negative urinary test result on a human chorionic gonadotropin pregnancy test on the day of randomization, before receiving any study product.
7. Males or females of childbearing potential who are using an effective birth control method recommended by the national health system for at least four (4) weeks before the first vaccination (for female participants only) and up to four (4) weeks after the third vaccination (i.e., for at least 4 months).

Exclusion Criteria:

1. Participant with major congenital abnormalities which in the opinion of investigator may affect the subject's participation in the study.
2. Participant concomitantly enrolled or scheduled to be enrolled in another trial.
3. Positive rapid test for HIV 1-2 confirmed by a positive blood test for human immunodeficiency virus (positive antibodies to HIV 1/2).
4. Participant seropositive for hepatitis B virus surface antigen (HBsAg).
5. Participant seropositive for hepatitis C virus (Antibodies to HCV).
6. Participant with active or chronic Schistosomiasis infection defined by a positive result for microscopy (Urine filtration, Kato-Katz (KK)) and point-of-care - circulating cathodic antigen (POC -CCA) and/or real-time PCR.
7. Participant with soiled transmitted helminths infections (STH) as diagnosed by microscopy (KK) and/or real-time PCR.
8. Participant with malaria infection/malaria as diagnosed by the blood smear.
9. Any other confirmed or suspected immunosuppressive or immunodeficient state such as asplenia, recurrent severe infections.
10. Body mass index (BMI) ≥ 35 kg/m2
11. Chronic use of systemic steroids (>2 mg/kg/day or >20 mg/day prednisolone equivalent for periods exceeding 10 days), cytotoxic or other immunosuppressive drugs.
12. Receipt of blood or blood-derived products in the past 3 months.
13. Participant who has received other vaccines 4 weeks prior to test vaccination or plans to receive any vaccine within 4 weeks of last dose of study vaccine, exception made for COVID-19 vaccines.
14. Known history of allergy to study vaccine components and/or excipients or other medications, or any other allergies deemed by the investigator to increase the risk of an adverse event if they were to participate in the trial.
15. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time resulting in contraindication for IM injections/blood extractions.
16. Any abnormality or chronic disease which in the opinion of the investigator might be detrimental for the safety of the participant and interfere with the assessment of the study objectives and compromise the health of the volunteers.
17. Any female participant who is lactating*, pregnant or planning for pregnancy** during the course of study period.
18. Individuals with behavioral or cognitive impairment or psychiatric disease or neural disorders that, in the opinion of the investigator, could interfere with the individual's ability to participate in the trial.
19. Any clinically significant abnormal finding on serum chemistry or hematology or urinalysis at the screening visit as per US FDA toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (any biological finding grade 4 constitutes an exclusion criteria).
20. Individuals who were research staff involved with the clinical study or family/household members of research staff.
21. As per Investigator's medical judgement individual could be excluded from the study despite meeting all inclusion/exclusion criteria mentioned above.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with of any Serious Adverse Events (SAEs)/ adverse events of special interest (AESI) from the time of the first study vaccination through the final study visit. | Day 1 through Day 224
Proportion of participants with immediate adverse events (reactogenicity events) within 60 min from the time of each study vaccination | Day 1 through Day 56
Proportion of participants with solicited local and solicited systemic AEs as measured for 7 days (inclusive) following immunization with the three different dose formulations. | Day 1 through Day 63
Proportion of participants with unsolicited AEs from the time of vaccination until 28 days post immunization with the three different dose formulations. | Day 1 through Day 84
Proportion of participants with clinical safety laboratory adverse events measured at 7 days and 28 days after each study vaccination. | Day 1 through Day 84

SECONDARY OUTCOMES:
For Sm-p80 IgG antibodies, seroconversion rate at approximately 4 weeks (28 days) after each dose of study vaccination as compared to baseline | Day 1 through Day 84
For Sm-p80 IgG antibodies, seroconversion rate at approximately 24 weeks after third dose of study vaccination as compared to baseline | Day 1 through Day 224
Geometric Mean Titers (GMTs) of serum Sm-p80 IgG antibodies at approximately 4 weeks after each dose of study vaccination. | Day 1 through Day 84
Geometric Mean Titers (GMTs) of serum Sm-p80 IgG antibodies at approximately 24 weeks after third dose of study vaccination. | Day 1 through Day 224

CONTACTS AND LOCATIONS:
Overall Officials: Florian Marks, Principal Investigator — International Vaccine Institute
Locations (2):
- Groupe de Recherche Action en Santé (GRAS), Ouagadougou, Burkina Faso
- Madagascar Institute for Vaccine Research (University of Antananarivo), Antananarivo, Madagascar

IPD SHARING:
Plan to Share IPD: No